CLINICAL TRIAL: NCT07290348
Title: Effect of Dynamic Hand Splint on Hand ROM Post Extensor Tendon Repair
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Magdy Helmi Mohamed Elmahdy Badra, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Magdy-MSc
Record Dates: First submitted 2025-12-05; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Splints; Range of Motion; Extensor Tendons of Finger Anomalies
MeSH Terms: conditions — Hapnes Boman Skeie syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dynamic hand splint (Experimental): This group included 20 patients suffering from cuts of the extensor tendon of their hand in zone 5 or 6 and underwent tendon repair surgery in this study. They wear a dynamic hand splint after 3 weeks post-operative for 2 months in addition to their conventional medical treatment and traditional care (dressing).
  Interventions: Other: customized dynamic hand splint; Other: traditional treatment (first stage); Other: traditional treatment (second and third stage)
- conventional medical treatment (Active Comparator): This group included 20 patients suffering from cuts of the extensor tendon of their hand in zone 5 or 6 and underwent tendon repair surgery in this study. They, without wearing a dynamic hand splint, received their conventional medical treatment and traditional care (dressing).
  Interventions: Other: traditional treatment (first stage); Other: traditional treatment (second and third stage)

INTERVENTIONS:
Other: customized dynamic hand splint — After 3 weeks of repair surgery, both groups were asked to take of the static splints, then the patients in group A (study group) were asked to wear customized dynamic hand splint daytime between sessions whole duration from third week post operative for 2 months till the end of the rehabilitation sessions, on the other hand the patients in group B (control group) were not asked to wear customized dynamic hand splint.
  Arms: dynamic hand splint
Other: traditional treatment (first stage) — All patients underwent a standardized rehabilitation program involving chair exercises. Key components included management of postoperative hand edema through distal-to-proximal massage to enhance tendon glide and range of motion; deep friction massage to reduce adhesions of postoperative scars; positive effects of massage therapy on hypertrophic and burn scar thickness; use of ultrasound on repaired tendons to minimize adhesions and promote healing; and gentle passive range of motion exercises for wrist and finger joints to gradually restore motion.
Other: traditional treatment (second and third stage) — This stage spanned two weeks following rehabilitation, during which all patients in both groups performed gentle stretching, active-assisted, and active free range of motion exercises to improve neuromuscular control and joint movements.
  This stage lasted one month, during which all patients engaged in active resisted range of motion, strengthening exercises, and functional training to restore muscle power and daily activity levels. Thera-band resistance training can improve muscle strength and functional fitness in older adults in community settings, serving as a safe and manageable physical activity that nursing staff can seamlessly integrate into daily routines.

SUMMARY:
The purpose of the study was to evaluate the effectiveness of dynamic hand splint on hand range of motion following extensor tendon repair.

DETAILED DESCRIPTION:
The extensor muscles to the digits are weaker; their capacity for work and their amplitude of glide are less than those of their flexor antagonists, yet they require a latitude of motion that is not necessary for flexor function. Extensor tendons are thinner and broader than flexor tendons. They are superficial in comparison with the flexor tendons, allowing adhesion to the fascial layers and skin. They have a broad tendon-to-bone interface that can result in dense adhesions. Shortening of the extensor tendon because of surgery may result in difficulty regaining full flexion. Dorsal swelling may prevent the tendons from gliding. Recreating the normal balance between intrinsic and extrinsic muscle/tendon units can be a challenging task for surgeons and therapists following extensor tendon injury. Common functional complications include loss of flexion, extensor lag, and decreased grip strength. To prevent these complications, extensor tendon approaches, similar to flexor tendon approaches, have evolved to include controlled passive and active mobilization using a dynamic splint immediately following surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients are both males and females.
* Their age will be in the range of 20-40 years.
* All patients suffering from extensor tendon injuries in zone 5 or 6.
* All patients undergo extensor tendon repair surgery.
* All patients will begin the treatment program from the third week post-operative.
* All patients enrolled in the study will have their informed consent.

Exclusion Criteria:

* The potential participants will be excluded if they meet one of the following criteria:
* Patients with associated diseases (diabetes mellitus, infectious diseases, autoimmune disease) that will interfere with the healing process.
* Patients taking medication that alters the healing process (e.g., corticosteroids, chemotherapy, or radiation).
* Pregnancy or epilepsy.
* Elderly patients.
* Skin disease.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2024-12-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
assessment of wrist range of motion | at baseline and after 1 months and 2 months
  The study measured the range of motion of the wrist at three stages: prior to treatment, after one month, and at the end of the treatment. Patients were positioned sitting with their elbows on a table.
  An electronic goniometer was employed for the measurements, ensuring the wrist was neutral (0°) for extension assessments. For wrist extension, the forearm was pronated and the elbow fully extended, with the goniometer aligned with the lateral side of the ulna and the fifth metacarpal for accurate measurement

SECONDARY OUTCOMES:
assessment of metacarpophalangeal joint range of motion | at baseline and after 1 months and 2 months
  The study measured the range of motion of the metacarpophalangeal joint of the fingers at three stages: prior to treatment, after one month, and at the end of the treatment.To measure the metacarpophalangeal joint, patients positioned their hands outside the table, while an electronic goniometer was aligned on the dorsal side of the metacarpal and proximal phalanx for accurate measurement.
assessment of interphalangeal joints' range of motion | at baseline and after 1 months and 2 months
  The study measured the range of motion of the proximal and distal interphalangeal joints of the fingers at three stages: prior to treatment, after one month, and at the end of the treatment.
  The measurement of proximal interphalangeal joints involved patients positioning their hands outside a table while an electronic goniometer was aligned on the dorsal side of the proximal and middle phalanx of the targeted finger. For Distal interphalangeal joints, the setup differed slightly, with alignment on the lateral side of the middle phalanx and distal phalanx of the targeted finger.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura international hospital, Dakahlia government, Egypt, Al Mansurah, Egypt